CLINICAL TRIAL: NCT03166943
Title: An Investigative Study on the Possible Effect of the Antiviral Inhibitors (Sofosbuvir and Daclatasvir) for Treatment of Hepatitis C Virus Infection in Cardiac Function
Brief Title: the Possible Effect of the Antiviral Inhibitors for Treatment of Hepatitis C Virus Infection in Cardiac Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rania Reda Yacoub, principal investigator, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SSD
Record Dates: First submitted 2017-05-11; First posted 2017-05-25 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Hepatitis
MeSH Terms: conditions — Hepatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Systolic function by echocardiography to100 Hepatitis C virus infected patients on continuous regimen ( sofosbuvir and daclatasvir )
  Interventions: Procedure: Systolic function by echocardiography
- Control group (Active Comparator): Diastolic function by echocardiography age and sex matched group of 30 patients with Hepatitis C virus who did not receive antiviral treatment ( sofosbuvir and daclatasvir )
  Interventions: Procedure: Diastolic function by echocardiography

INTERVENTIONS:
Procedure: Systolic function by echocardiography — Echocardiography for evaluation of systolic function:
  * by biplane Simpson's method.
  * by speckle tracking:
  Arms: study group
Procedure: Diastolic function by echocardiography — Echocardiography for evaluation of diastolic function:
  * Left atrial Volume
  * Mitral Inflow Patterns
    * Pulsed wave Doppler
    * Mitral inflow patterns include normal, impaired left ventricular relaxation, pseudonormal, and restrictive left ventricular filling patterns.
  * Tissue Doppler Annular Early and Late Diastolic Velocities
    * Pulsed wave tissue doppler imaging
    * Primary measurements include the systolic , early diastolic, and late diastolic velocities.
  Arms: Control group

SUMMARY:
It has been known for many years that the heart and the liver are intimately related. There is a mutual interaction between the function of the heart and the liver and a broad spectrum of acute and chronic entities that affect both the heart and the liver. Chronic hepatitis C virus infection affects more than 3% (170 million) of the world's population.

DETAILED DESCRIPTION:
Assessment of systolic function by echocardiography will be done to 100 hepatitis C virus infected patients who receive antiviral treatment (sofosbuvir and daclatasvir) by biplane simpson's method and by speckle tracking.

Assessment of diastolic function by echocardiography to 30 hepatitis C virus infected patients who will not receive antiviral treatment, by left atrium volume , mitral inflow pattern , tissue doppler annular early and late diastolic velocities .

ELIGIBILITY:
Inclusion Criteria:

1. patients on continuous regimen (Sofosbuvir and daclatasvir) for 3 months
2. normal baseline trans thoracic echocardiography
3. normal Electrocardiography

Exclusion Criteria:

1 - Diabetes mellitus, hypertension and chronic kidney disease. 2- Hepatitis C virus patients with any baseline Electrocardiography abnormality.

3- Patients with underlying any structural heart disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2017-05-10 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with ventricular dysfunction | 3 months
  The percentage of ventricular dysfunction in hepatitis C virus patients who received antiviral treatment in comparison with patients with hepatitis C virus who didn't receive antiviral treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No